CLINICAL TRIAL: NCT01916850
Title: A Phase 1b, Single-center, Double-blind, Randomized, Placebo-controlled Study on the Safety, Tolerability, and Pharmacokinetic Effects of Multiple Doses of LX4211 400 mg qd and LX4211 800 mg qd in Healthy Subjects
Brief Title: Study to Determine the Safety, Tolerability and Pharmacokinetics Following Multiple Doses of LX4211 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX4211.1-110-NRM; LX4211.110 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2013-07-29; First posted 2013-08-06 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
MeSH Terms: interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- LX4211 Low Dose (Experimental): 400 mg of LX4211 administered once daily for 10 consecutive days
  Interventions: Drug: LX4211 400 mg
- LX4211 High Dose (Experimental): 800 mg of LX4211 administered once daily for 10 consecutive days
  Interventions: Drug: LX4211 800 mg
- Placebo (Placebo Comparator): Identical placebo administered once daily for 10 consecutive days
  Interventions: Drug: LX4211 Placebo

INTERVENTIONS:
Drug: LX4211 400 mg
  Arms: LX4211 Low Dose
Drug: LX4211 800 mg
  Arms: LX4211 High Dose
Drug: LX4211 Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of multiple oral doses of LX4211 400 mg and LX4211 800 mg (administered once daily for 10 consecutive days) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ≥ 18 to ≤ 55 years of age
* Vital signs at Screening in the following ranges: systolic blood pressure, 90-140 mm Hg; diastolic blood pressure, 50-90 mm Hg; heart rate, 50-100 bpm
* Body mass index (BMI) ≥18 and ≤35 kg/sq m
* Willing and able to provide written informed consent

Exclusion Criteria:

* Use of any medication (prescription, over-the-counter, herbal tea, or supplements) within 5 days of dosing
* Use of any investigational agent or study treatment within 30 days of dosing
* Use of any protein or antibody-based therapeutic agents within 3 months of Screening
* Prior exposure to LX4211
* Use of cigarettes or any tobacco products within 2 months prior to Screening and while participating in the study
* History of bariatric surgery or any other gastrointestinal surgery that may induce malabsorption
* History of any major surgery within 6 months of Screening
* History of any hypersensitivity to the inactive components of LX4211
* History of renal disease or significantly abnormal kidney function tests
* History of hepatic disease or significantly abnormal liver function tests
* History of any active infection within 14 days prior to Day 1
* History of alcohol or substance abuse within 2 years prior to Day 1
* Donation or loss of >400 mL of blood or blood product within 3 months of dosing
* Positive urine glucose at Screening
* Positive urine screen for drugs of abuse, or urine test for alcohol at Screening or Day -1
* Inability or difficulty swallowing pills
* Unable or unwilling to communicate or cooperate with the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to Day 10

SECONDARY OUTCOMES:
Area under the curve | Days 1 through 10

CONTACTS AND LOCATIONS:
Overall Officials: Ikenna (Ike) Ogbaa, M.D., Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, Dallas, Texas, United States